CLINICAL TRIAL: NCT01080963
Title: Prospective Randomised Study of Daptomycin as Antibiotic Prophylaxis of Sternal Wound Infections After Median Sternotomy
Brief Title: Daptomycin as Antibiotic Prophylaxis of Sternal Wound Infections
Acronym: DaPro
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Martin Strueber, Martin Strueber, MD, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCBC134ADAPRO; 2007-004611-61 (EudraCT Number)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Wound Infection
Keywords: Prophylaxis; Antibiotic; Sternotomy; Heart-Lung Machine
MeSH Terms: conditions — Wound Infection | interventions — Daptomycin; Cefuroxime

ARMS (2):
- Daptomycin (Active Comparator)
  Interventions: Drug: Daptomycin
- Cefuroxime (Active Comparator)
  Interventions: Drug: Cefuroxime

INTERVENTIONS:
Drug: Daptomycin — one infusion of 350 mg intraoperatively after disconnection from the heart-lung machine as an add-on to standard antibiotic prophylaxis
  Other Names: Cubicin
  Arms: Daptomycin
Drug: Cefuroxime — 1500 mg intravenous 30min preoperatively during anesthesia and 1500 mg intravenous intraoperatively after disconnection from the heart-lung machine
  Arms: Cefuroxime

SUMMARY:
The purpose of this study is to show that the incidence of sternal wound infections at day 30 after cardiac surgery is 50% lower with the additional use of Daptomycin on top of a standard antibiotic prophylaxis as compared to the standard antibiotic prophylaxis alone.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-80
* written informed consent (IC)

Exclusion Criteria:

* pregnant and lactating women
* patients operated for a transplantation
* patients with a increased myopathy risk
* patients with a creatinine clearance < 30ml/min; patients on hemodialysis
* patients after a previous sternotomy
* treatment with any antibiotics 14 days prior study start
* treatment with Daptomycin or Cefuroxime within 3 month prior study start

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2008-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Incidence of sternal wound infection is at least 50% lower if Daptomycin is used on top of a standard antibiotic prophylaxis as compared to the standard antibiotic prophylaxis alone | day 30

SECONDARY OUTCOMES:
Incidence of sternal wound infections at day 30 after cardiac surgery | day 30

CONTACTS AND LOCATIONS:
Overall Officials: Martin Strueber, Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Department of Cardiothoracic, Transplant and Vascular surgery, Hanover, Germany